CLINICAL TRIAL: NCT02793908
Title: The Role of the Subcutaneous Progesterone in Luteal Phase Supplementation in Patients With Endometriosis
Brief Title: Subcutaneous Progesterone Supplementation in Patients With Endometriosis
Acronym: PleyrisEndom
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Fulvio Zullo, Full Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMagnaGraecia
Record Dates: First submitted 2016-06-02; First posted 2016-06-08 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Endometriosis
Keywords: Endometriosis; Subcutaneous progesterone; luteal phase
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pleyris (Experimental): Subcutaneous progesterone will be administered 25 mg a day from the day following the ovulation for 14 days
  Interventions: Drug: Pleyris
- Crinone8 (Active Comparator): Vaginal progesterone will be administered 90 mg a day from the day following the ovulation for 14 days
  Interventions: Drug: Crinone8

INTERVENTIONS:
Drug: Pleyris — Luteal phase will be supplemented starting by the ovulation day for 14 days
  Other Names: Subcutaneous progesterone
  Arms: Pleyris
Drug: Crinone8 — Luteal phase will be supplemented starting by the ovulation day for 14 days
  Other Names: vaginal progesterone
  Arms: Crinone8

SUMMARY:
The aim of the study protocol will be to compare the efficacy of subcutaneous progesterone (25 mg / day; Pleyris, IBSA Institut Biochimique SA) with vaginal progesterone (90 mg / day; Crinone, Merck Serono) administered during the luteal phase in term of pelvic pain reduction in patients with grade I-II endometriosis and / or endometrioma <4 cm subjected to time intercourses or COS/IUI cycles.

DETAILED DESCRIPTION:
Patients with grade I-II endometriosis and / or endometrioma <4 cm subjected to time intercourses or COS/IUI cycles will be subjected to subcutaneous or vaginal progesterone for their luteal phase supplementation in time intercourses or IUI cycles.

The aim of the study protocol will be to compare the efficacy of subcutaneous progesterone (25 mg / day; Pleyris, IBSA Institut Biochimique SA) with vaginal progesterone (90 mg / day; Crinone, Merck Serono) administered during the luteal phase in term of pelvic pain reduction

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic or ultrasonographic diagnosis of endometriosis grade I-II and / or endometrioma <4 cm;
* Menstrual VAS score> 5 cm before the last menstrual period with progesterone treatment
* Infertility for at least 1 year
* Body Mass Index 19 to 30 kg / m2
* Basal FSH serum <15 IU / ml
* Normal levels of serum prolactin
* Normal uterine cavity and fallopian patency

Exclusion Criteria:

* Previous ovarian surgery
* Endocrine disorders (eg polycystic ovary syndrome, thyroid disease, hyperprolactinemia, hypogonadotropic hypogonadism)
* Reduced ovarian reserve (basal levels of FSH> 15 IU / mL)
* Acute or chronic infectious state
* Chronic drug intake, alcohol, or drugs that affect cognitive functions, alertness and / or mood
* Psychiatric disorders
* Kidney or liver diseases
* Male factor infertility

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Delta VAS pain | 7 days after the end of the menstrual period subsequent to the luteal supplementation
  Patients will be asked to score their menstrual pain using a VAS scale

SECONDARY OUTCOMES:
Analgesic use | 7 days after the end of the menstrual period subsequent to the luteal supplementation
  Patients will be asked how many vials of analgesics they needed during their menstrual period
Pregnancy rate | 30 days after the end of the menstrual period subsequent to the luteal supplementation
  The percentage of pregnancies achieved in both arms will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Fulvio Zullo, Study Director — Magna Graecia University of Catanzaro; Roberta Venturella, Principal Investigator — Magna Graecia University of Catanzaro
Locations (1):
- Magna Graecia University - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro, CZ, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be published at the end of the study.